CLINICAL TRIAL: NCT00039741
Title: A Phase II/III Randomized, Open-Label Study of Combination Antiretroviral Regimens and Treatment-Switching Strategies in HIV-1-Infected Antiretroviral Naive Children Between 30 Days and 18 Years of Age
Brief Title: Anti-HIV Drug Regimens and Treatment-Switching Guidelines in HIV Infected Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); PENTA Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P390; PENPACT-1B; 10106 (Registry Identifier: DAIDS ES); PENTA 9/PACTG 390
Record Dates: First submitted 2002-06-07; First posted 2002-06-11 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Viral Load; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Racivir; Stavudine; efavirenz; Nevirapine; CDP-Diacylglycerol-Inositol 3-Phosphatidyltransferase; Adenosine Monophosphate; Indinavir; Nelfinavir; Saquinavir; Ritonavir

ARMS (4):
- PI/1K (Experimental): Two NRTIs plus a PI with a regimen change recommended at when viral load reaches 1000 copies/ml or higher
  Interventions: Drug: NRTIs (ABC, FTC, FTC/TDF, 3TC, 3TC/AZT, d4T, TDF, ddC, AZT); Drug: PIs (AMP, IDV, LPV/r, NFV, SQV, RTV)
- NNRTI/1K (Experimental): 2 NRTIs plus an NNRTI with a regimen change recommended when viral load reaches 1,000 copies/ml or higher
  Interventions: Drug: NRTIs (ABC, FTC, FTC/TDF, 3TC, 3TC/AZT, d4T, TDF, ddC, AZT); Drug: NNRTIs (EFV, NVP)
- PI/30K (Experimental): 2 NRTIs plus 1 PI with a regimen change recommended when viral load reaches 30,000 copies/ml or higher
  Interventions: Drug: NRTIs (ABC, FTC, FTC/TDF, 3TC, 3TC/AZT, d4T, TDF, ddC, AZT); Drug: PIs (AMP, IDV, LPV/r, NFV, SQV, RTV)
- NNRTI/30K (Experimental): 2 NRTIs plus an NNRTI with a regimen change recommended when viral load reaches 30,000 copies/ml or higher
  Interventions: Drug: NRTIs (ABC, FTC, FTC/TDF, 3TC, 3TC/AZT, d4T, TDF, ddC, AZT); Drug: NNRTIs (EFV, NVP)

INTERVENTIONS:
Drug: NRTIs (ABC, FTC, FTC/TDF, 3TC, 3TC/AZT, d4T, TDF, ddC, AZT) — Accepted NRTIs: abacavir sulfate (ABC), emtricitabine (FTC), emtricitabine/Tenofovir disoproxil fumarate (FTC/TDF), lamivudine (3TC), lamivudine/zidovudine (3TC/AZT), stavudine (d4T), tenofovir disoproxil fumarate (TDF), zalcitabine (ddC), zidovudine (AZT) Prescribed per participant's doctor
  Other Names: 2 NRTIs/PI, change@viral load 1000 copies/ml or higher; 2 NRTIs/PI, change@viral load 30,000 copies/ml or higher; 2 NRTIs/NNRTI, change@viral load 1000 copies/ml or higher; 2 NRTIs/NNRTI, change@viral load 30,000 copies/ml or higher
Drug: NNRTIs (EFV, NVP) — Accepted NNRTIs: efavirenz (EFV), nevirapine (NVP)
  Prescribed per participant's doctor
  Other Names: 2 NRTIs/NNRTI, change@viral load 1000 copies/ml or higher; 2 NRTIs/NNRTI, change@viral load 30,000 copies/ml or higher
  Arms: NNRTI/1K; NNRTI/30K
Drug: PIs (AMP, IDV, LPV/r, NFV, SQV, RTV) — Accepted PIs: amprenavir (APV). indinavir sulfate (IDV), lopinavir/ritonavir (LPV/r), nelfinavir mesylate (NFV), saquinavir (SQV), ritonavir (RTV)
  Prescribed per participant's doctor
  Other Names: 2 NRTIs/PI, change@viral load 1000 copies/ml or higher; 2 NRTIs/PI, change@viral load 30,000 copies/ml or higher
  Arms: PI/1K; PI/30K

SUMMARY:
Little is known about what treatment combinations are best for HIV infected children. This study examined the long-term effectiveness of different anti-HIV drug combinations in children and strategies for switching treatment if the first treatment does not work. The study enrolled children who had not previously taken anti-HIV medication. Participants in this study were recruited in the United States, South America and Europe.

Some European children may also enroll in a substudy that will observe changes in body fat in children taking anti-HIV medications.

DETAILED DESCRIPTION:
Antiretroviral therapy in children aims to prolong clinical and immunologic health. Currently, there are no data defining a particular highly active antiretroviral therapy (HAART) strategy as the optimal first-line therapy for children. This study evaluated the long-term efficacy of two HAART regimens used as initial therapy: 1) two nucleoside reverse transcriptase inhibitors (NRTIs) plus a protease inhibitor (PI), and 2) two NRTIs plus a nonnucleoside reverse transcriptase inhibitor (NNRTI). It also evaluated different strategies for switching therapy when the initial regimen fails. The long-term nature of this study should clarify whether early switching of therapy improves immunologic and virologic outcomes, or results in a more rapid exhaustion of treatment options. The study was conducted in the United States and in Europe.

Participants in this study had a CD4 cell count and viral load test during a screening visit. Participants had an entry visit that included blood and urine tests. Participants were then randomly assigned to one of four groups: Groups PI/1K and PI/30K received two NRTIs plus a PI; Groups NNRTI/1K and NNRTI/30K received two NRTIs plus an NNRTI. The medications allowed in the study were: abacavir, didanosine, emtricitabine, emtricitabine/tenofovir disoproxil fumarate, lamivudine, lamivudine/zidovudine, stavudine, tenofovir disoproxil fumarate, zalcitabine, and zidovudine (NRTIs); efavirenz and nevirapine (NNRTIs); efavirenz/emtricitabine/tenofovir disoproxil fumurate (NNRTI/NRTI); and amprenavir,atazanavir, darunavir, fosamprenavir calcium, indinavir, lopinavir/ritonavir, nelfinavir, saquinavir, ritonavir, and tipranavir (PIs). Note: Per the 06/28/05 amendment of this trial, emtricitabine, emtricitabine/tenofovir disoproxil fumarate, and tenofovir dioproxil fumarate were added to the list of medications that could be included in a participant's treatment regimen.

For participants whose initial regimen failed, or who experienced clinical disease progression (indicated by the development of a new CDC Category C diagnosis) or other clinical disease progression at or after Week 24 of first-line therapy, second-line therapy was strongly encouraged. (However, if poor adherence was suspected as a possible reason for an increase in HIV viral load, the site and the clinician were to try to improve patient adherence and obtain additional confirmatory viral load values within a five-week time frame.) In second-line therapy, participants who initially took NRTIs with a PI switched to NRTIs and an NNRTI. Participants who initially took NRTIs and an NNRTI switched to NRTIs and a PI. The timing of the switch was based on the participant's group: Groups PI/1K and NNRTI/1K switched to second-line treatment when viral load was 1,000 copies/ml or greater; Groups PI/30K and NNRTI/30K switched to second-line treatment when viral load was 30,000 copies/ml or greater. Participants who failed second-line therapy discontinued study treatment and were offered the best available therapy at the discretion of the clinician.

Participants had study visits at Weeks 2, 4, 8, 12, 16, 24, and every 12 weeks thereafter until the drug regimen was switched to second-line treatment. Participants then had a re-entry visit and the schedule of visits restarted. Participants were in the study between 4 and 7 years, depending on when they enrolled. All study visits included medical history, a physical exam, and blood collection. Urine collection occurred at most visits. Participants were asked to complete adherence questionnaires and PACTG participants underwent neuropsychological assessments at selected visits.

All participants in this study were encouraged to coenroll in PACTG 219C, Long-Term Effects of HIV Exposure and Infection in Children. Participants in the European portion of the study may be asked to enroll in a substudy to observe the development and progression of lipodystrophy syndrome in children.

ELIGIBILITY:
Inclusion Criteria:

* Older than 30 days and younger than 18 years of age (may enroll up to the day before their 18th birthday)
* HIV infected
* Not previously on HAART or received anti-HIV drugs for less than 56 consecutive days after birth to prevent mother-to-infant HIV transmission. Participants who have previously received nevirapine for the prevention of mother-to-infant HIV transmission are not eligible for this study.
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Grade 3 or 4 clinical or laboratory toxicity. More information on this criterion can be found in the protocol.
* Active opportunistic infection or a serious bacterial infection at the time of study entry
* Pancreas, nervous system, blood, liver, or kidney problems that make it impossible to take study medications
* Taking any medication that cannot be combined with the study medications in first-line therapy
* Received therapy for cancer
* Pregnant or breastfeeding

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 266 (Actual)
Dates: Start 2002-08; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross E. McKinney, Jr., MD, Study Chair — Duke University; Ann J. Melvin, MD, Study Chair — Division of Infectious Diseases, Children's Hospital and Medical Center, Seattle, WA
Locations (31):
- United States (29):
  - Usc La Nichd Crs, Alhambra, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - Children's Hospital of Los Angeles NICHD CRS, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Connecticut Children's Med. Ctr., Hartford, Connecticut
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - UMDNJ - Robert Wood Johnson Med. School, Div. of Allergy, Immunology & Infectious Diseases, New Brunswick, New Jersey
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - Oregon Health & Science Univ. - Dept. of Peds., Div. of Infectious Disease, Portland, Oregon
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas
  - Seattle Children's Hospital CRS, Seattle, Washington
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Brogly S, Williams P, Seage GR 3rd, Oleske JM, Van Dyke R, McIntosh K; PACTG 219C Team. Antiretroviral treatment in pediatric HIV infection in the United States: from clinical trials to clinical practice. JAMA. 2005 May 11;293(18):2213-20. doi: 10.1001/jama.293.18.2213. PMID 15886376
- [Background] Havens PL. Principles of antiretroviral treatment of children and adolescents with human immunodeficiency virus infection. Semin Pediatr Infect Dis. 2003 Oct;14(4):269-85. doi: 10.1053/j.spid.2003.09.005. PMID 14724792
- [Background] Hoody DW, Fletcher CV. Pharmacology considerations for antiretroviral therapy in human immunodeficiency virus (HIV)-infected children. Semin Pediatr Infect Dis. 2003 Oct;14(4):286-94. doi: 10.1053/j.spid.2003.09.004. PMID 14724793
- [Background] McKinney RE Jr, Cunningham CK. Newer treatments for HIV in children. Curr Opin Pediatr. 2004 Feb;16(1):76-9. doi: 10.1097/00008480-200402000-00014. PMID 14758118
- [Result] PENPACT-1 (PENTA 9/PACTG 390) Study Team; Babiker A, Castro nee Green H, Compagnucci A, Fiscus S, Giaquinto C, Gibb DM, Harper L, Harrison L, Hughes M, McKinney R, Melvin A, Mofenson L, Saidi Y, Smith ME, Tudor-Williams G, Walker AS. First-line antiretroviral therapy with a protease inhibitor versus non-nucleoside reverse transcriptase inhibitor and switch at higher versus low viral load in HIV-infected children: an open-label, randomised phase 2/3 trial. Lancet Infect Dis. 2011 Apr;11(4):273-83. doi: 10.1016/S1473-3099(10)70313-3. Epub 2011 Jan 31. PMID 21288774
- See also: Click here for more information about ACTG 219C (NCT00006304) — http://www.clinicaltrials.gov/ct/show/NCT00006304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at Pediatric AIDS Clinical Trials Group (PACTG) units in the U.S. and Puerto Rico, and Paediatric European Network for Treatment of AIDS (PENTA) units in Argentina, Austria, the Bahamas, Brazil, France, Germany, Italy, Romania, Spain, the United Kingdom and Ireland. Enrollment started 9/25/02 and ended 9/7/05.
Pre-assignment Details: Participants were stratified by age (<3 years versus 3+ years), origin (PACTG site or PENTA site), and exposure versus no exposure to antiretroviral therapy perinatally. 266 children were randomized, of whom 3 are excluded from all analyses (2 had consent withdrawn by parents after randomization, 1 was ineligible).
Groups:
- PI/1K: Two nucleoside reverse transcriptase inhibitors (NRTI) plus a protease inhibitor (PI)with a regimen change recommended when viral load is 1000 copies/ml or higher
- NNRTI/1K: 2 NRTIs plus a nonnucleoside reverse transcriptase inhibitor (NNRTI) with a regimen change recommended when viral load reaches 1,000 copies/ml or higher
- PI/30K: Two NRTIs plus a PIwith a regimen change recommended when viral load is 30,000 copies/ml or higher
Period: Overall Study
Arm/Group | PI/1K | NNRTI/1K | PI/30K | NNRTI/30K
Started | 66 | 68 | 65 | 64
Death | 0 | 1 | 0 | 0
Completed | 51 | 56 | 54 | 50
Not Completed | 15 | 12 | 11 | 14
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 5 | 2
Not completed — Confounding medical condition | 1 | 0 | 0 | 0
Not completed — Not able to get to clinic | 5 | 2 | 0 | 3
Not completed — Moved | 3 | 2 | 3 | 6
Not completed — Non-compliance with protocol | 1 | 0 | 1 | 0
Not completed — Withdrew consent | 0 | 5 | 0 | 1
Not completed — Missed final visit | 2 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PI/1K | NNRTI/1K | PI/30K | NNRTI/30K | Total
Number analyzed (Participants) | 66 | 68 | 65 | 64 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (5.7) | 7.0 (5.4) | 7.9 (5.4) | 6.9 (5.0) | 7.5 (5.4)
Age, Customized [Number; unit: participants]
  >30 days to <=12 months | 10 | 12 | 7 | 11 | 40
  >12 months to <=3 years | 8 | 7 | 8 | 5 | 28
  >3 to <=9 years | 19 | 27 | 24 | 29 | 99
  >9 to <=14 years | 14 | 13 | 13 | 10 | 50
  >14 years to <18 years | 15 | 9 | 13 | 9 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 32 | 32 | 127
  Male | 36 | 35 | 33 | 32 | 136
Region of Enrollment [Number; unit: participants] — Sites in the US and Puerto Rico were enrolled through PACTG, and other sites were enrolled through PENTA
  participants
    United States | 18 | 20 | 16 | 18 | 72
    Puerto Rico | 1 | 1 | 1 | 0 | 3
    Argentina | 1 | 4 | 3 | 3 | 11
    Austria | 1 | 0 | 0 | 1 | 2
    Bahamas | 2 | 0 | 2 | 0 | 4
    Brazil | 12 | 11 | 9 | 9 | 41
    France | 3 | 3 | 5 | 6 | 17
    Germany | 5 | 6 | 3 | 7 | 21
    Italy | 7 | 4 | 5 | 6 | 22
    Romania | 8 | 7 | 9 | 7 | 31
    Spain | 1 | 0 | 1 | 0 | 2
    United Kingdom | 7 | 11 | 9 | 6 | 33
    Ireland | 0 | 1 | 2 | 1 | 4
Viral Load [Mean (Standard Deviation); unit: Log10 copies/ml] — Log10 HIV-1 RNA (copies/ml)
  Log10 copies/ml | 5.2 (0.8) | 5.0 (0.8) | 5.0 (0.8) | 5.1 (0.8) | 5.1 (0.8)
PENTA/PACTG site [Number; unit: participants]
  PENTA | 47 | 47 | 48 | 46 | 188
  PACTG | 19 | 21 | 17 | 18 | 75
CD4 percent (percentage of total lymphocytes that are CD4 cells) [Mean (Standard Deviation); unit: CD4%] | 18 (12) | 18 (10) | 18 (11) | 17 (12) | 18 (11)

OUTCOME MEASURES:

1. Primary Outcome: Change in Viral Load Measured in log10 HIV-1 RNA Copies/ml
Time Frame: Baseline visit and 4 years after Study Entry
Population: Intent-to-treat analyses for those subjects who had data at baseline and 4 years. Analyses were done by collapsing groups to examine drug class (regardless of switch point) and switch point (regardless of drug class).
Measure: Mean (Standard Error); unit: log10 HIV-1 RNA
Groups:
- Drug Class/PI: Participants randomized to receive a PI-based regimen, regardless of switch point.
- Drug Class/NNRTI: Participants randomized to receive an NNRTI-based regimen, regardless of switch point.
- Switch Point (1K): Participants randomized to switch to second-line therapy when HIV-1 RNA is >=1,000 copies/mL, regardless of drug class.
- Switch Point (30K): Participants randomized to switch to second-line therapy when HIV-1 RNA is >=30,000 copies/mL, regardless of drug class.
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 118 | 116 | 117 | 117
log10 HIV-1 RNA | -3.16 (0.09) | -3.31 (0.09) | -3.26 (0.09) | -3.20 (0.09)
Statistical Analysis 1: Comparison: Drug Class/PI vs Drug Class/NNRTI; Test type: Superiority or Other; p = 0.26, Interval regression; Adjusted for baseline HIV-1 RNA, age (<3 years vs 3 years), origin (PACTG vs PENTA sites), and perinatal ART exposure versus no exposure; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.41 to 0.11], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Switch Point (1K) vs Switch Point (30K); Test type: Superiority or Other; p = 0.56, Interval regression; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.20 to 0.32], Standard Error of Mean 0.13

2. Secondary Outcome: Rate of Grade 3 or Higher Signs, Symptoms, or Laboratory Abnormalities Experienced
Description: Adverse events were graded according to the following guidelines:
  PACTG: "The Manual for Expedited Reporting of Adverse Events to DAIDS" (DAIDS EAE Manual) dated May 6, 2004.
  PENTA: International Conference for Harmonization (ICH) requirements and the EU Clinical Trials Directive 2001/20/EC (20).
  A rating of Grade 3 is severe and Grade 4 is life-threatening. The rate of serious (Grade 3 or above)events is reported as the number of events per 100 child/years.
Time Frame: Up to 6 yrs. (average 4.85 yrs.)
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: events/100 child-years
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 131 | 132 | 134 | 129
events/100 child-years | 0.16 [0.08 to 0.31] | 0.17 [0.09 to 0.31] | 0.16 [0.08 to 0.31] | 0.17 [0.09 to 0.31]

3. Secondary Outcome: Participants With Significant HIV-related Clinical Events, Defined as CDC Category C (AIDS Defining) Diagnoses (Except for Recurrent Bacterial Infections)or Death
Time Frame: Up to 6 yrs. (average 4.85 yrs.)
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 131 | 132 | 134 | 129
participants | 6 | 4 | 5 | 5

4. Secondary Outcome: Time to Switching to an Alternative Class ART Regimen (Based on Initial Randomized Regimen)
Description: 25th Percentiles in weeks from randomization to starting an alternative class ART regimen (based on initial randomized regimen)
Time Frame: Up to 6 yrs. (average 4.85 yrs.)
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Weeks (25th Percentile)
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 131 | 132 | 134 | 129
Weeks (25th Percentile) | NA [295 to NA] — Fewer than 50% of participants reached the switching criteria, so the median and 75th percentile are undefined. | NA [142 to NA] — Fewer than 50% of participants reached the switching criteria, so the median and 75th percentile are undefined. | NA [142 to NA] — Fewer than 50% of participants reached the switching criteria, so the median and 75th percentile are undefined. | NA [240 to NA] — Fewer than 50% of participants reached the switching criteria, so the median and 75th percentile are undefined.

5. Secondary Outcome: Time to HIV-1 RNA of 400 Copies/ml or Greater During First-line Therapy or Permanent Discontinuation of First-line Therapy
Description: 25th Percentiles in weeks from randomization HIV-1 RNA of 400 copies/ml or greater during first-line therapy or permanent discontinuation of first-line therapy.
Time Frame: Up to 6 yrs. (average 4.85 yrs.)
Population: Intent to treat
Measure: Number; unit: Weeks (25th Percentile)
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 131 | 132 | 134 | 129
Weeks (25th Percentile) | 36 | 68 | 41 | 72

6. Secondary Outcome: Time to HIV-1 RNA of 30,000 Copies/ml or Greater During Second-line Therapy or Permanent Discontinuation of Second-line Therapy
Description: 25th Percentiles in weeks from randomization to HIV-1 RNA of 30,000 copies/ml or greater during second-line therapy or permanent discontinuation of second-line therapy
Time Frame: Up to 6 yrs. (average 4.85 yrs.)
Population: Intent to treat
Measure: Number; unit: Weeks (25th Percentile)
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 28 | 32 | 37 | 23
Weeks (25th Percentile) | 126 | 267 | 267 | 228

7. Secondary Outcome: Number of Children With an HIV-1 RNA Level Less Than 400 Copies/ml Regardless of Therapy at Week 204
Time Frame: Week 204
Population: Intent to treat. Numbers are reported among participants who had an HIV-1 RNA value and were in follow-up at week 204.
Measure: Number; unit: participants
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 112 | 114 | 114 | 112
participants | 92 | 93 | 95 | 90

8. Secondary Outcome: Change in CD4% From Randomization to 4 Years
Time Frame: Randomization to 4 years
Population: Intent to treat, for participants who had CD4% values available at 4 years and at baseline.
Measure: Mean (Standard Deviation); unit: CD4 percent (% of total lymphocytes)
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 131 | 132 | 134 | 129
CD4 percent (% of total lymphocytes) | 13.7 (0.8) | 15.2 (0.8) | 15.1 (0.8) | 13.9 (0.8)

9. Secondary Outcome: Number of Children With HIV-1 RNA Less Than 400 Copies/ml and on Original Randomized Therapy at 24 Weeks
Time Frame: 24 weeks
Population: Intent to treat - numbers are reported among participants who had an HIV-1 RNA value and were in follow-up at week 24.
Measure: Number; unit: participants
Arm/Group | Drug Class/PI | Drug Class/NNRTI | Switch Point (1K) | Switch Point (30K)
Number analyzed (Participants) | 130 | 129 | 132 | 127
participants | 92 | 98 | 99 | 91

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 6.8 years, with a median of 5 years. The last study visit was August 31, 2009. ICH (International Conference for Harmonization) criteria were used for determining Serious Adverse Events.
Description: Only events with Grade 3 or greater are reported. No Other (Non-Serious) Adverse events occurred with 5% or greater frequency.
Arm/Group | PI/1K | NNRTI/1K | PI/30K | NNRTI/30K
Serious Adverse Events (participants affected / at risk) | 9/66 | 10/68 | 14/65 | 15/64
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68 | 0/65 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PI/1K (N=66) | NNRTI/1K (N=68) | PI/30K (N=65) | NNRTI/30K (N=64)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anemia megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aplastic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Progressive external ophthalmoplegia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea, viral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema nodosum (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Appendicitis, perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis, viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis, viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphkinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup, infectious (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No